CLINICAL TRIAL: NCT04363255
Title: Efficacy and Safety of First-line Etoposide/Platinum-based Chemotherapy Followed by Toripalimab Combined With Anlotinib for Maintenance in Extensive Small Cell Lung Cancer: A Single-arm, Multicentral Phase II Study
Brief Title: First-line Chemotherapy Followed by Toripalimab Combined With Anlotinib for Maintenance in ES-SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, The head of radiotherapy department in Taizhou Hospital, Taizhou Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LDQ-202004
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Carboplatin; Cisplatin; toripalimab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maintenance group (Experimental): After 4-6 cycles of EP/EC chemotherapy regiment, maintenance therapy with toripalimab and anlotinib was followed and continued until disease progression.
  Interventions: Drug: Etoposide Injection; Drug: Carboplatin Injection; Drug: Cisplatin injection; Drug: Toripalimab; Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Etoposide Injection — Etoposide(100mg/m2, d1-3, q3w) combined with platinum was the first-line chemotherapy in 4-6 cycles, and then JS001 combined with anlotinib as maintenance therapy were followed.
  Other Names: Etoposide
Drug: Carboplatin Injection — Carboplatin(AUC 5, d1, q3w) or Cisplatin combined with etoposide was the first-line chemotherapy in 4-6 cycles, and then JS001 combined with anlotinib as maintenance therapy were followed.
  Other Names: Carboplatin
Drug: Cisplatin injection — Cisplatin(75mg/m2, d1, q3w) or carboplatin combined with etoposide was the first-line chemotherapy in 4-6 cycles, and then JS001 combined with anlotinib as maintenance therapy were followed.
  Other Names: Cisplatin
Drug: Toripalimab — After 4-6 cycles of chemotherapy, JS001(240mg, d1, q3w) combined with anlotinib were followed and continued until disease progression.
  Other Names: JS001
Drug: Anlotinib hydrochloride — After 4-6 cycles of chemotherapy, anlotinib(12mg qd, d1-14, q3w) combined with JS001 were followed and continued until disease progression.
  Other Names: Anlotinib

SUMMARY:
Our aim in this study was to evaluate the efficacy and safety of etoposide combined with cisplatin or carboplatin (EC/EP) chemotherapy regimens followed by toripalimab combined with anlotinib for maintenance in extensive small cell lung cancer(ES-SCLC).

DETAILED DESCRIPTION:
Lung cancer is the most leading malignant tumor, among which small cell lung cancer accounts for about 15%. Approximately 65% of new patients were diagnosed with ES-SCLC at the first visit with less than 6 months of median PFS (mPFS) and 8-13 months of median OS (mOS). Platinum combined with etoposide or irinotecan chemotherapy is the first-line standard chemotherapy treatment. Despite high objective response of initial treatment, it is evitable to develop chemotherapy resistance and the effects of follow-up line treatment is dissatisfying. Therefore, combination therapy may be promising and efficient.

Anlotinib, the brand new multi-target protein tyrosine kinase (PTK) blockers, could normalize distribution of blood vessels in the tumor, gather T cells and enhance effect of immune drugs via vascular endothelial growth factor receptor (VEGFR), platelet-derived growth factor receptor (PDGFR), fibroblast growth factor receptor (FGFR), type Ⅲ tyrosine kinase and others signal pathways, and then inhibit the growth, proliferation and differentiation of lung cancer cells. According to ALTER1202 study, anlotinib played a promising role in local tumor control and effectively prolonged PFS in third line or more for ES-SCLC patients. Meanwhile, immunocheckpoint inhibitors can improve tumor immune microenvironment, relieve VEGF-mediated immunosuppression, reduce Treg activity, promote tumor antigen presenting ability and better infiltrate T cell into the tumor to play an anti-tumor effect. Emerging studies have shown that immunocheckpoint inhibitors, such as Atezolizumab, Pembrolizumab and Nivolumab, can effectively improve ORR, DoR and survival in SCLC patients. In terms of molecular mechanisms, immunocheckpoint inhibitors and vascular targeting drugs complemented and the combination of two drugs has superior efficacy in non-small cell lung cancer (NSCLC), just as it shown in IMpower150 and other studies. However, the role of immunocheckpoint inhibitors in maintenance therapy in SCLC were disappointing in CheckMate451 and a study of pembrolizumab, although it obtained some victories in first line or more for SCLC.

In summary, the investigators proposed that first-line etoposide/platinum-based chemotherapy followed by toripalimab combined with anlotinib for maintenance may prolong chemo-resistance in extensive small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must sign a specific informed consent form prior to clinical trial; 2. Extensive stage small cell lung cancer confirmed by histology or cytology; 3. Patients did not receive any system treatment before or only received EP/EC chemotherapy (time from the last medication of chemotherapy to the beginning of maintenance treatment must be ≤21 days); 4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1; 5. An estimated survival duration of >5 months from the beginning of chemotherapy; 6. Age no less than 18; 7. A measurable lesion on image; 8. Patients with asymptomatic brain metastases or symptomatic brain metastases which were stable after treatment; 9. Before the first dose of drugs for study, patients should have appropriate organ function and the laboratory results must meet conditions as following: Blood routine examination: neutrophil absolute value (ANC) ≥1.5×109/L, platelet (PLT) ≥100×109/L, hemoglobin content (HGB) ≥9g/dl; Adequate hepatic function: bilirubin ≤1.5×ULN mg/dl, creatinine clearance ≥ 50 ml/min; Adequate hepatic function: Aspartate aminotransferase (AST) /alanine aminotransferase (ALT)> 2.5 × upper limit of normal (ULN) or > 5 × ULN (patients with liver metastasis), alkaline phosphatase (ALP) ≤2.5×ULN or ≤5×ULN (patients with bone metastasis), Total bilirubin (TB) ≤1.5×ULN, albumin (ALB)>30g/dl; Coagulation function: international normalized ratio (INR) ≤1.5×ULN, activated partial thromboplastin time (APTT) ≤1.5×ULN; Urine routine: 24-hour urine protein<1g (if urine protein ≥2+, additional 24-hour urine protein is required); Others: serum lipase or amylase ≤1.5×ULN or >1.5×ULN (subjects clinically or radiologically diagnosed with pancreatitis).

Exclusion Criteria:

* 1. Patients received EP/EC regiment received the last medication ≥21 days before maintenance treatment, or received other systematic anti-tumor treatment for ES-SCLC; 2. Patients with epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) mutation; 3. Patients received any other experimental drugs or participated in another interventional clinical study within 4 weeks prior to signing the informed consent; 4. Patients received other systemic or local antitumor therapy (including but not limited to the use of other drugs for SCLC maintenance therapy or radiotherapy, but CR/PR subjects are allowed to use prophylactic cranial irradiation (PCI) after induction period treatment); 5. Patients with active and untreated brain metastases or carcinoma meningitis in CT or MRI examination during screening stage; 6. Patients with other malignant tumors within 5 years, except for curable malignant tumors (carcinoma in situ or stage I tumor), such as cervical carcinoma in situ, basal cell or squamous cell skin cancer and so on); 7. Patients received corticosteroids (>10mg/ day methyl prednisolone or equivalent dose) or other immunosuppressants (inhalation or local use of steroids and adrenal replacement treatment were permitted in the absence of an active autoimmune disease) less than 14 days prior to maintenance medications; 8. Patients with chronic or acute active hepatitis B (HBsAg positive and hepatitis B virus (HBV) DNA copy number >ULN), or HCV positive (HCV Ab positive and HCV RNA positive); Hepatitis B patients with previous HBV infection or who have been cured (HBsAg negative, HBcAb positive and HBV DNA copy number < ULN) were allowed to be enrolled; 9. Patients with interstitial lung disease, drug-induced pneumonia, radiation pneumonitis requiring steroid treatment, or active pneumonia with clinical symptoms; or other lung diseases causing moderate or severe lung dysfunction; Active pulmonary tuberculosis or the need for anti-tuberculosis treatment; 10. Patients who were allergy to one of research drugs, or allergy to any one of the immunocheckpoint inhibitors or other platinum; 11. Female patients during pregnant and lactation period, or patients were plan to pregnant; 12. Patients with factors that may cause the study to be forced to terminate halfway according to investigators' judgement, such as poor compliance, other serious diseases requiring combined treatment and so on.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Duration of time from the start of chemotherapy to the time of disease progression, assessed up to 3 years
  PFS
Overall survival (OS) | Duration of time from the start of chemotherapy to the time of outcome events, assessed up to 3 years
  OS

SECONDARY OUTCOMES:
Adverse event (AE) | Duration of time from the start of treatment to the end of study, assessed up to 3 years
  The acute and chronic AE profiles associated with the study regimen using CTCAE v5.0
Objective response rate (ORR) | Duration of time from the start of treatment to the end of study, assessed up to 3 years
  ORR was the sum percentage of partial response (PR) and stable disease (SD) according to RECIST v1.1
Disease control rate (DCR) | Duration of time from the start of treatment to the end of study, assessed up to 3 years
  DCR was the sum percentage of complete response (CR), partial response (PR) and stable disease (SD) according to RECIST v1.1
Duration of response (DoR) | Duration of time from the start of treatment response to the time of disease progression, assessed up to 3 years
  DoR

CONTACTS AND LOCATIONS:
Overall Officials: Dongqing Lv, MD, Principal Investigator — Enze Hospital affiliated Taizhou hospital of Wenzhou Medical University
Locations (2):
- China (2):
  - Enze Hospital, affiliated Taizhou Hospital of Wenzhou Medical University, Taizhou, Zhejiang
  - Haihua, Yang, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
make individual participant data (IPD) available